CLINICAL TRIAL: NCT05832333
Title: Post-marketing Surveillance Study for the Use of VaxigripTetra®, a Quadrivalent Influenza Vaccine Administered Via Intramuscular Route in Subjects Aged 6 to 35 Months in Republic of Korea
Brief Title: Postmarketing Surveillance Study for Quadrivalent Influenza Vaccine (VaxigripTetra®) in Subjects Aged 6 to 35 Months
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: GQM00015
Record Dates: First submitted 2023-04-11; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: VaxigripTetra® — Suspension for injection Injection intramuscular
  Other Names: Quadrivalent influenza vaccine (split-virion, inactivated) - QIV

SUMMARY:
Multi-center, observational, active safety surveillance study in participants aged 6 to 35 months in Korea under routine clinical practices.

DETAILED DESCRIPTION:
The planned duration of each participant's participation in the study will be 21 to 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 35 months on the day of enrolment
* Informed consent form has been signed and dated by the parent or other legally acceptable representative
* Receipt of one dose of VaxigripTetra® on the day of inclusion in routine practice according to the approved local product insert

Exclusion Criteria:

- Participation at the time of study enrolment (or in the 4 weeks preceding the enrolment) or planned participation during the present study period in a clinical study investigating a vaccine, drug, medical device, or medical procedure

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants aged 6 to 35 months will be enrolled after receipt of one dose of VaxigripTetra® during a routine health care visit.
  Participants will be enrolled on the day of vaccination (first or second vaccination) and will be followed-up for only one vaccination.
  Planned number of subjects: 670 subjects aged 6 to 35 months Planned number of country: 1 (Republic of Korea) Planned number of sites: 12
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Occurence of solicited injection site or systemic reactions | Up to 7 days after vaccination
  Percentage of participants reporting
  * injection site reactions: pain, erythema, swelling, induration, ecchymosis
  * systemic reactions for infants and toddlers ≤ 23 months: fever, vomiting ,crying abnormal, drowsiness, appetite lost, irritability
  * systemic reactions for children aged 2 to 3 years: fever, headache, malaise, myalgia, shivering
Occurence of unsolicited adverse events (AEs) | Up to 21(+7) days after vaccination
  Percentage of participants with unsolicited (spontaneously reported) injection site reactions occurring within 28 days after each injection and unsolicited systemic AEs between each injection and up to 28 days after the last injection
Occurrence of serious adverse events (SAEs) throughout the study participation | Up to 21(+7) days after vaccination
  Percentage of participants with SAEs, including AESIs, throughout the study

CONTACTS AND LOCATIONS:
Locations (12):
- South Korea (12):
  - Site 003, Gangwon-do
  - Site 002, Gwangju
  - Site 004, Gyeonggi-do
  - Site 005, Gyeonggi-do
  - Site 008, Gyeonggi-do
  - Site 011, Gyeonggi-do
  - Site 015, Gyeonggi-do
  - Site 006, Gyeongsangnam-do
  - Site 010, Gyeongsangnam-do
  - Site 009, Seoul
  - Site 012, Seoul
  - Site 014, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://www.vivli.org